CLINICAL TRIAL: NCT04044911
Title: Randomised Controlled Trial of a Task Model Approach (CogWatch) to Tea Making Training in Stroke Apraxia and Action Disorganisation Syndrome
Brief Title: Trial Using CogWatch for Tea Making Training in Stroke Apraxia and Action Disorganisation Syndrome
Acronym: CogWatchTea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ERN_12-0683B
Record Dates: First submitted 2019-07-05; First posted 2019-08-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-03

CONDITIONS: Stroke; Apraxias
Keywords: Activity of daily living; Stroke; Apraxia; Action of daily living; Cup of tea
MeSH Terms: conditions — Stroke; Apraxias

STUDY DESIGN:
Intervention Model Description: Crossover randomized control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tea making followed by stepping (Active Comparator): Five 1-hour weekly tea making training sessions in which progress is monitored and feedback given using a computer-based system that implements a Markov Decision Process (MDP) task model (CogWatch) is followed after a 3-week break by a control condition in which participants receive five 1-hour weekly stepping training sessions.
  Interventions: Behavioral: Task model (CogWatch)
- Stepping followed by tea making (Active Comparator): A control condition comprising five 1-hour weekly stepping training sessions is followed after a 3-week break by five 1-hour weekly tea making training sessions in which progress is monitored and feedback given using a computer-based system that implements a Markov Decision Process (MDP) task model (COgWatch)
  Interventions: Behavioral: Task model (CogWatch)

INTERVENTIONS:
Behavioral: Task model (CogWatch)

SUMMARY:
Apraxia and action disorganization syndrome after stroke can disrupt activities of daily living (ADL). Occupational therapy has been effective in improving ADL performance, however, inclusion of multiple tasks means it is unclear which therapy elements contribute to improvement. This study evaluates the efficacy of a task model approach to ADL rehabilitation, comparing training in making a cup of tea with a gait training control condition.

DETAILED DESCRIPTION:
Apraxia and action disorganization syndrome (AADS) after stroke can disrupt activities of daily living (ADLs). Occupational therapy has been effective in improving ADL performance, however, inclusion of multiple tasks means it is unclear which therapy elements contribute to improvement.

This trial evaluates the efficacy of a task model approach to ADL rehabilitation, comparing training in making a cup of tea with a stepping training control condition.

Stroke survivors with AADS participate in a cross-over randomized controlled study. Participants attend five 1-hour tea making training sessions in which progress is monitored and feedback given using a computer-based system which implements a Markov Decision Process (MDP) task model (CogWatch). In a control condition participants receive five 1-hour stepping sessions.

Analysis compares tea making training with stepping training effects on error reduction and time taken in making 4 different tea types. A complex tea preparation task (making two different cups of tea simultaneously) is used to test for generalisation of training effects.

ELIGIBILITY:
Inclusion Criteria:

* greater than 2 months post stroke; medically stable; failing at least one of four praxis items in the Birmingham Cognitive Screen (BCoS) or a document filing task.

Exclusion Criteria:

* recent stroke (less than 2 months post stroke); not medically stable

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2014-12-04 (Actual); Study Completion 2014-12-04 (Actual)

PRIMARY OUTCOMES:
Change in tea making accuracy | 3 assessments over 12 weeks
  In three assessment sessions (initial, post-phase 1 training, post-phase 2 training), participants are seated at a table with objects and ingredients required for making a cup of tea placed in standard positions. Participants are instructed to make 8 cups of tea, one at a time, comprising two of each of the following; black tea, black tea with sugar, tea with milk and tea with milk and sugar. Each trial is recorded with a video camera.
  Videos of the participants making simple tea are analysed by a researcher blinded to the session definition. The summed errors across the 8 tea making trials at each assessment are used to provide a measure of accuracy for each participant.
  Change in tea making accuracy pre- and post-training of tea making is contrasted with change in tea making accuracy pre- and post-training of stepping.
Change in tea making speed | 3 assessments over 12 weeks
  In three assessment sessions (initial, post-phase 1 training, post-phase 2 training), participants are seated at a table with objects and ingredients required for making a cup of tea placed in standard positions. Participants are instructed to make 8 cups of tea, one at a time, comprising two of each of the following; black tea, black tea with sugar, tea with milk and tea with milk and sugar. Each trial is recorded with a video camera.
  Videos of the participants making simple tea are analysed by a researcher blinded to the session definition. The average completion time is used as a measure of speed for each participant.
  Change in tea making speed pre- and post-training of tea making is contrasted with change in tea making speed pre- and post-training of stepping.

SECONDARY OUTCOMES:
Tea making accuracy at follow-up | 2 assessments over 15 weeks
  In a fourth, follow-up assessment session (7 or 15 weeks post-tea making training), participants are seated at a table with objects and ingredients required for making a cup of tea placed in standard positions. Participants are instructed to make 8 cups of tea, one at a time, comprising two of each of the following; black tea, black tea with sugar, tea with milk and tea with milk and sugar. Each trial is recorded with a video camera.
  Videos of the participants making simple tea are analysed by a researcher blinded to the session definition. The summed errors across the 8 tea making trials at each assessment are used to provide a measure of accuracy for each participant.
  Tea making accuracy at follow-up is compared with tea making accuracy post-training of tea making.
Change in complex tea making accuracy | 3 assessments over 12 weeks
  In three assessment sessions (initial, post-phase 1 training, post-phase 2 training), participants are seated at a table with objects and ingredients required for making two cups of tea placed in standard positions. Participants are instructed to make 4 cups of tea, two at a time, comprising one cup with tea, lemon and 1 sugar cube and the other with tea, milk and 2 sweeteners. Each trial is recorded with a video camera.
  Videos of the participants making complex tea are analysed by a researcher blinded to the session definition. The summed errors across the 4 tea making trials at each assessment are used to provide a measure of accuracy for each participant.
  Change in complex tea making accuracy pre- and post-training of tea making is contrasted with change in complex tea making accuracy pre- and post-training of stepping.

CONTACTS AND LOCATIONS:
Overall Officials: Alan M WIng, PhD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howe J, Chua W, Sumner E, Drozdowska B, Laverick R, Bevins RL, Jean-Baptiste E, Russell M, Rotshtein P, Wing AM. The efficacy of a task model approach to ADL rehabilitation in stroke apraxia and action disorganisation syndrome: A randomised controlled trial. PLoS One. 2022 Mar 3;17(3):e0264678. doi: 10.1371/journal.pone.0264678. eCollection 2022. PMID 35239707